CLINICAL TRIAL: NCT02687542
Title: A 15-WEEK, PHASE 2, DOUBLE BLIND, RANDOMIZED, PLACEBO-CONTROLLED, DOSE RANGING STUDY TO INVESTIGATE THE EFFICACY, SAFETY AND TOLERABILITY OF PF-06649751 IN SUBJECTS WITH MOTOR FLUCTUATIONS DUE TO PARKINSON'S DISEASE
Brief Title: Efficacy, Safety and Tolerability of PF-06649751 in Parkinson's Disease Patients With Motor Fluctuations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated 25Sep17 due to insufficient efficacy. Not due to safety reasons.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: B7601003; 2015-004912-39 (EudraCT Number); A-ROSE PD (Other: Alias Study Number); A-ROSE (Other: Alias Study Number)
Record Dates: First submitted 2016-01-29; First posted 2016-02-22 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Motor Fluctuation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PF-06649751 low dose (1 mg QD) (Experimental): PF-06649751 low dose level (1 mg QD)
  Interventions: Drug: PF-06649751 low dose (1 mg QD)
- PF-06649751 middle dose 1 (3 mg QD) (Experimental): PF-06649751 lower middle dose 1 (3 mg QD)
  Interventions: Drug: PF-06649751 middle dose 1 (3 mg QD)
- PF-06649751 middle dose 2 (7 mg QD) (Experimental): PF-06649751 higher middle dose 2 (7 mg QD)
  Interventions: Drug: PF-06649751 middle dose 2 (7 mg QD)
- PF-06649751 high dose (15 mg QD) (Experimental): PF-06649751 high dose (15 mg QD)
  Interventions: Drug: PF-06649751 high dose (15 mg QD)

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-06649751 low dose (1 mg QD) — PF-06649751 low dose (1 mg QD)
  Arms: PF-06649751 low dose (1 mg QD)
Drug: PF-06649751 middle dose 1 (3 mg QD) — PF-06649751 lower middle dose 1 (3 mg QD)
  Arms: PF-06649751 middle dose 1 (3 mg QD)
Drug: PF-06649751 middle dose 2 (7 mg QD) — PF-06649751higher middle dose 2 (7 mg QD)
  Arms: PF-06649751 middle dose 2 (7 mg QD)
Drug: PF-06649751 high dose (15 mg QD) — PF-06649751 high dose (15 mg QD)
  Arms: PF-06649751 high dose (15 mg QD)

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of PF-06649751 in Parkinson's disease patients who experience motor-fluctuations.

DETAILED DESCRIPTION:
The study has a randomized, double-blind, placebo-controlled parallel group design. Approximately 198 subjects will be randomized to 5 treatment groups. Each subject will participate in the study for approximately 23 weeks including a 30 day screening period, 15 week double blind treatment period, and an approximately 28 day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential and/or male subjects between the ages of 40 and 85 years, inclusive.
* Clinical diagnosis of Parkinson's disease.
* Able to refrain from any Parkinson's disease medication not permitted by the protocol.

Exclusion Criteria:

* Female of childbearing potential
* History or presence of atypical Parkinsonian syndrome.
* History of surgical intervention for Parkinson's disease.
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality.
* Any condition possibly affecting drug absorption.
* Participation in other studies involving investigational drug(s), or treatment with any investigational drug within 30 days.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (33):
  - Xenoscience, Inc, Phoenix, Arizona
  - St Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arcadia Neurology Center, Arcadia, California
  - Faculty Physicians and Surgeons of Loma Linda University School of Medicine, Loma Linda, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Hoag Memorial Hospital, Newport Beach, California
  - SC3 Research Group, Inc, Pasadena, California
  - Neurosearch-Torrance, Torrance, California
  - Associated Neurologists of Southern Connecticut, PC, Fairfield, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - University of South Florida, Tampa, Florida
  - Vero Beach Neurology and Research Institute, Vero Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - CRI Worldwide, LLC, Marlton, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Dent Neurosciences Research Center ,Inc. DBA Dent Neurologic Institute, Amherst, New York
  - Dent Neurologic Institute, Orchard Park, New York
  - Duke University Medical center, Durham, North Carolina
  - Duke University/Duke Neurology/Department of Neurology, Durham, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Abington Neurological Associates, Ltd., Willow Grove, Pennsylvania
  - Rhode Island Hospital/ Brown University Medical School, Providence, Rhode Island
  - AS Clinical Research Consultants of North Texas, PLLC, Greenville, Texas
  - Baylor College of Medicine, Houston, Texas
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
- Canada (2):
  - Montreal Neurological Hospital Research Pharmacy, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- France (6):
  - CHU de Grenoble Alpes, Grenoble
  - CHU de Grenoble Alpes, La Tronche
  - CHRU de Lille-Hopital Roger Salengro, Lille
  - Hopital de la Timone APHM, Marseille
  - Hopital de La Timone, Marseille
  - Hopital La Pitie-Salpetriere, Paris
- Germany (5):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - St. Josef-Hospital GmbH, Bochum
  - Universitaetsklinikum Carl Gustav Carus Klinik und Poliklinik fur Neurologie, Dresden
  - Klinikum rechts der Isar der Technischen Universitaet Muenchen, München
  - Universitaetsklinik Ulm, Ulm
- Japan (5):
  - Asahikawa Medical center, Asahikawa, Hokkaido
  - Medical Corporation Abe Neurology Clinic, Morioka, Iwate
  - Tazuke Kofukai Medical Research Institute Kitano Hospital, Kita-ku, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
- Spain (6):
  - Hospital Clinico Universitario, Santiago de Compostela, A Coruna
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Policlinica de Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario y Politecnico la Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7601003

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The participants swallowed 3 tablets once daily (QD) at approximately the same time each morning within approximately 5 minutes without being manipulated or chewed prior to being swallowed.
  Duration of treatment was 15 weeks. A follow-up visit was at Week 17, 2 weeks after discontinuation of Placebo. A follow-up phone visit was scheduled at Week 19 for participant's safety.
- PF-06649751 1 mg QD; PF-06649751 3 mg QD; PF-06649751 7 mg QD; PF-06649751 15 mg QD: The participants swallowed 3 tablets QD at approximately the same time each morning within approximately 5 minutes without being manipulated or chewed prior to being swallowed.
  Duration of treatment was 15 weeks including: 3-week titration of PF-06649751 administered QD to the randomized target dose; 2-week stabilization period for dose adjustment after reaching the target dose; 5-week Period A of PF-06649751 administered QD adjunctive to stable doses of L-Dopa; 5-week Period B (maintenance period) of PF-06649751 administered QD adjunctive to stable doses of L-Dopa.
  A follow-up visit was at Week 17, 2 weeks after discontinuation of PF-06649751. A follow-up phone visit was scheduled at Week 19 for participant's safety.
Period: Overall Study
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Started | 23 | 13 | 15 | 13 | 44
Completed | 15 | 1 | 1 | 3 | 24
Not Completed | 8 | 12 | 14 | 10 | 20
Not completed — Medication error without associated AEs | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Other | 5 | 9 | 10 | 6 | 5
Not completed — Adverse Event | 3 | 1 | 3 | 2 | 9
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD | Total
Number analyzed (Participants) | 23 | 13 | 15 | 13 | 44 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.04 (8.79) | 66.92 (8.79) | 63.80 (7.76) | 67.77 (9.36) | 63.41 (8.47) | 64.97 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 4 | 18 | 40
  Male | 17 | 7 | 9 | 9 | 26 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 1 | 1 | 3 | 11
  Not Hispanic or Latino | 20 | 10 | 13 | 12 | 40 | 95
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 2 | 1 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 2 | 1 | 6
  White | 20 | 12 | 12 | 9 | 36 | 89
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily OFF Time at Week 10
Description: A paper Hauser diary was utilized to record motor state for half-hour intervals. Participants completed the diary by answering whether they had been OFF for 3 consecutive days in the week prior to each visit (except Day 28 visit), including 3 consecutive days during the week prior to Day 0 (Randomization).
  The daily OFF time was calculated as the average of the 3 consecutive daily OFF hours from the Hauser diary at each visit.
Time Frame: Week 10; Baseline was defined as the average daily OFF time (using 3 Hauser patient diary days) prior to Day -1 (study derived day and equalled to nominal visit day 0).
Population: Full Analysis Set consisted of all participants randomized who completed at least 1 post-dose efficacy measurement (Hauser home diary).
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 21 | 7 | 9 | 9 | 41
Hours | -0.969 (0.4092) | -1.173 (0.3482) | -1.316 (0.3289) | -1.480 (0.3460) | -1.663 (0.4297)
Statistical Analysis 1: Comparison: Placebo vs PF-06649751 15 mg QD; Test type: Other — Bayesian Dose Response Analysis; p = 0.5776, Bayesian Dose Response Analysis — Bayesian Predictive Test for Emax (the additive increase over Placebo in the response of PF-06649751 at a theoretically infinite dose) Monotonicity; Estimate and 90% credible interval of Bayesian dose response difference from placebo; Bayesian Dose Reponse Estimate = -0.693, 90% CI 2-sided [-1.713 to 0.304], Standard Error of Mean 0.6162

2. Secondary Outcome: Change From Baseline in Daily OFF Time
Description: A paper Hauser diary was utilized to record motor state for half hour intervals. Participants completed the diary by answering whether they had been OFF for 3 consecutive days in the week prior to each visit (except Day 28 visit), including 3 consecutive days during the week prior to Day 0 (Randomization).
  The daily OFF time was calculated as the average of the 3 consecutive daily OFF hours from the Hauser diary at each visit.
  Results at Week 15 should be interpreted with caution given almost half the participants were not available for this analysis at Week 15 as compared to Week 10 and the complicated nature of protocol changes that impacted the study design after Week 10.
Time Frame: Weeks 3, 5, 10 and 15; Baseline was defined as the average daily OFF time (using 3 Hauser patient diary days) prior to Day -1 (study derived day and equalled to nominal visit day 0).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 21 | 7 | 9 | 9 | 41
Hours
  Change at Week 3: number analyzed (Participants) | 18 | 6 | 8 | 6 | 37
  Change at Week 3 | -0.67 (0.620) | -0.82 (1.237) | -0.55 (1.091) | -1.82 (1.182) | -1.01 (0.464)
  Change at Week 5: number analyzed (Participants) | 17 | 5 | 6 | 7 | 32
  Change at Week 5 | -0.63 (0.490) | -2.04 (1.054) | -2.23 (0.964) | -1.41 (0.937) | -1.24 (0.392)
  Change at Week 10: number analyzed (Participants) | 16 | 3 | 2 | 5 | 25
  Change at Week 10 | -0.99 (0.628) | -0.60 (1.423) | -1.00 (1.508) | -2.07 (1.187) | -1.63 (0.502)
  Change at Week 15: number analyzed (Participants) | 7 | 1 | 1 | 3 | 14
  Change at Week 15 | 1.05 (1.063) | -0.67 (2.960) | -2.75 (2.936) | -1.09 (1.687) | -2.47 (0.793)

3. Secondary Outcome: Change From Baseline in Daily ON Time With Troublesome Dyskinesia
Description: A paper Hauser diary was utilized to record motor state for half hour intervals. The participants answered the Hauser diary on whether they had been ON with troublesome dyskinesia. A diary day started with the interval 24:00-0:30 through 23:30-24:00 on each chronological day for 3 consecutive days. On the days recording the home diary, participants made an entry every 30 minutes during their normal waking time and upon awakening from time asleep.
  The daily ON hours was calculated as the average of the 3 consecutive daily ON hours from the Hauser diary at each visit.
  Results at Week 15 should be interpreted with caution given almost half the participants were not available for this analysis at Week 15 as compared to Week 10 and the complicated nature of protocol changes that impacted the study design after Week 10.
Time Frame: Weeks 3, 5, 10 and 15; Baseline was defined as the average daily ON time with Troublesome Dyskinesia (using 3 Hauser patient diary Days) prior to Day -1 (study derived day and equalled to nominal visit Day 0).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 21 | 7 | 9 | 9 | 41
Hours
  Change at Week 3: number analyzed (Participants) | 18 | 6 | 8 | 6 | 37
  Change at Week 3 | 0.17 (0.236) | 0.07 (0.467) | 0.19 (0.417) | 0.01 (0.464) | 0.23 (0.179)
  Change at Week 5: number analyzed (Participants) | 17 | 5 | 6 | 7 | 32
  Change at Week 5 | 0.23 (0.198) | -0.21 (0.415) | -0.02 (0.388) | 0.45 (0.363) | 0.03 (0.162)
  Change at Week 10: number analyzed (Participants) | 16 | 3 | 2 | 5 | 25
  Change at Week 10 | 0.13 (0.191) | 0.24 (0.464) | 0.32 (0.529) | -0.39 (0.389) | 0.13 (0.167)
  Change at Week 15: number analyzed (Participants) | 7 | 1 | 1 | 3 | 14
  Change at Week 15 | 0.01 (0.642) | -0.43 (1.349) | -0.29 (1.263) | 0.54 (1.071) | -0.21 (0.463)

4. Secondary Outcome: Change From Baseline in Daily ON Time Without Troublesome Dyskinesia
Description: A paper Hauser diary was utilized to record motor state for half hour intervals. The participants answered the Hauser diary on whether they had been ON without troublesome dyskinesia. A diary day started with the interval 24:00-0:30 through 23:30-24:00 on each chronological day for 3 consecutive days. On the days recording the home diary, participants made an entry every 30 minutes during their normal waking time and upon awakening from time asleep.
  The daily ON hours was calculated as the average of the 3 consecutive daily ON hours from the Hauser diary at each visit.
  Results at Week 15 should be interpreted with caution given almost half the participants were not available for this analysis at Week 15 as compared to Week 10 and the complicated nature of protocol changes that impacted the study design after Week 10.
Time Frame: Weeks 3, 5, 10 and 15; Baseline was defined as the average daily ON time without Troublesome Dyskinesia (using 3 Hauser patient diary days) prior to Day -1 (study derived day and equalled to nominal visit Day 0)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 21 | 7 | 9 | 9 | 41
Hours
  Change at Week 3: number analyzed (Participants) | 18 | 6 | 8 | 6 | 37
  Change at Week 3 | 0.61 (0.577) | 1.74 (1.173) | -0.49 (1.047) | 1.93 (1.128) | 0.77 (0.443)
  Change at Week 5: number analyzed (Participants) | 17 | 5 | 6 | 7 | 32
  Change at Week 5 | 0.02 (0.548) | 2.39 (1.150) | 1.31 (1.058) | 1.12 (1.029) | 1.31 (0.436)
  Change at Week 10: number analyzed (Participants) | 16 | 3 | 2 | 5 | 25
  Change at Week 10 | 0.61 (0.618) | 0.92 (1.413) | 0.45 (1.598) | 2.64 (1.194) | 1.65 (0.508)
  Change at Week 15: number analyzed (Participants) | 7 | 1 | 1 | 3 | 14
  Change at Week 15 | -0.81 (1.099) | 0.37 (2.999) | -4.48 (3.192) | 0.94 (1.781) | 1.50 (0.825)

5. Secondary Outcome: Change From Baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III
Description: MDS-UPDRS Part III assessed the motor signs of Parkinson's disease and was administered by the investigator. It was comprised of 33 sub-scores based on 18 items, several with right, left or other body distribution scores. Each question was anchored with 5 responses that were linked to commonly accepted clinical terms: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. If more than 7 of the Part III items were missing, the score for that time point was missing, otherwise MDS-UPDRS Part III score was imputed as sum of the non-missing items*(total number of items)/ (number of items non-missing). The MDS-UPDRS Part III total score range is 0-132. Higher score indicated more severe motor signs of Parkinson's disease.
  Results at Week 15 should be interpreted with caution given almost half the participants were not available for this analysis at Week 15 as compared to Week 10 and the complicated nature of protocol changes that impacted the study design after Week 10.
Time Frame: Weeks 1, 2, 3, 4, 5, 10 and 15; Baseline was defined as the Day -1 (study derived day and equalled to nominal visit Day 0) measurement
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 21 | 7 | 9 | 9 | 41
units on a scale
  Change at Week 1 | -3.90 (2.054) | -4.44 (3.965) | -4.61 (3.593) | -1.90 (3.594) | -3.22 (1.524)
  Change at Week 2: number analyzed (Participants) | 11 | 1 | 0 | 1 | 20
  Change at Week 2 | -0.95 (2.078) | -15.78 (6.252) |  | 0.56 (6.129) | -3.70 (1.584)
  Change at Week 3: number analyzed (Participants) | 10 | 1 | 0 | 0 | 20
  Change at Week 3 | -3.80 (2.848) | -12.39 (8.240) |  |  | -3.06 (2.069)
  Change at Week 4: number analyzed (Participants) | 18 | 7 | 9 | 9 | 37
  Change at Week 4 | -6.28 (2.182) | -0.84 (3.940) | -2.48 (3.572) | -2.91 (3.575) | -6.05 (1.574)
  Change at Week 5: number analyzed (Participants) | 18 | 6 | 6 | 8 | 34
  Change at Week 5 | -5.12 (2.386) | -6.14 (4.414) | 3.10 (4.347) | -1.22 (3.935) | -4.86 (1.765)
  Change at Week 10: number analyzed (Participants) | 17 | 5 | 2 | 6 | 30
  Change at Week 10 | -5.09 (1.967) | -2.21 (3.902) | 5.77 (5.365) | -2.36 (3.607) | -9.32 (1.526)
  Change at Week 15: number analyzed (Participants) | 8 | 1 | 1 | 3 | 15
  Change at Week 15 | -0.18 (3.170) | 7.72 (8.660) | 2.09 (9.495) | -5.44 (5.364) | -1.84 (2.519)

6. Secondary Outcome: Change From Baseline in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I, II, IV, and Total Score
Description: Each question of Part I,II or IV with 5 responses was linked to the same clinical terms as Part III.The score was missing if more than 7 items were missing for a time point; otherwise Part I,II or IV score was imputed as sum of non-missing items*(total number of items)/(number of items non-missing).•PartI (Non-Motor Aspects of Experiences of Daily Living) assessed non-motor experiences of daily living using 13questions(Range:0-52).•PartII(Motor Aspects of Experiences of Daily Living) assessed motor experiences of daily living using 13questions(Range:0-52).•PartIV(Motor Complications) assessed motor complications,dyskinesias, and motor fluctuations using historical and objective information with 6questions(Range:0-24).•MDS-UPDRS Total Score:the sum of Parts I,II,III,and IV(Range:0-260).Higher score indicated more severe motor signs of Parkinson's disease.Week15's results were interpreted cautiously given almost half participants were not available for the analysis as compared to Week10
Time Frame: Weeks 5, 10 and 15; Baseline was defined as the Day -1 (study derived day and equalled to nominal visit Day 0) measurement
Population: Full Analysis Set included all participants randomized who completed at least 1 postdose efficacy measurement(Hauser home diary).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 21 | 7 | 9 | 9 | 41
units on a scale
  Change at Week 5 (Part I Score): number analyzed (Participants) | 16 | 6 | 6 | 8 | 34
  Change at Week 5 (Part I Score) | -0.75 (5.508) | -0.83 (1.941) | 0.67 (4.885) | 2.00 (4.408) | 1.12 (4.879)
  Change at Week 10 (Part I Score): number analyzed (Participants) | 16 | 5 | 2 | 6 | 30
  Change at Week 10 (Part I Score) | -0.69 (4.557) | -0.80 (2.168) | -1.00 (2.828) | 0.00 (2.449) | 0.17 (4.086)
  Change at Week 15 (Part I Score): number analyzed (Participants) | 7 | 1 | 1 | 3 | 15
  Change at Week 15 (Part I Score) | -2.86 (6.176) | 2.00 (NA) — Only 1 participant evaluable in this treatment group. | 6.00 (NA) — Only 1 participant evaluable in this treatment group. | -1.00 (1.732) | 1.00 (5.745)
  Change at Week 5 (Part II Score): number analyzed (Participants) | 18 | 6 | 6 | 8 | 34
  Change at Week 5 (Part II Score) | 0.06 (5.836) | -1.83 (2.639) | 3.00 (4.940) | -0.03 (3.083) | -0.24 (4.068)
  Change at Week 10 (Part II Score): number analyzed (Participants) | 17 | 5 | 2 | 6 | 30
  Change at Week 10 (Part II Score) | -0.35 (5.267) | -1.00 (1.225) | 5.00 (1.414) | 0.13 (2.428) | -0.43 (4.240)
  Change at Week 15 (Part II Score): number analyzed (Participants) | 8 | 1 | 1 | 3 | 15
  Change at Week 15 (Part II Score) | -1.38 (4.779) | 2.00 (NA) — Only 1 participant evaluable in this treatment group. | 8.00 (NA) — Only 1 participant evaluable in this treatment group. | -2.42 (5.270) | 1.47 (5.986)
  Change at Week 5 (Part IV Score): number analyzed (Participants) | 18 | 6 | 6 | 8 | 34
  Change at Week 5 (Part IV Score) | -1.50 (2.895) | -0.83 (2.401) | -0.50 (4.848) | 0.25 (2.053) | -0.65 (2.806)
  Change at Week 10 (Part IV Score): number analyzed (Participants) | 17 | 5 | 2 | 6 | 30
  Change at Week 10 (Part IV Score) | -2.00 (2.318) | 0.80 (1.304) | -3.00 (5.657) | 0.00 (1.789) | -1.13 (3.530)
  Change at Week 15 (Part IV Score): number analyzed (Participants) | 8 | 1 | 1 | 3 | 15
  Change at Week 15 (Part IV Score) | -2.75 (2.493) | -2.00 (NA) — Only 1 participant evaluable in this treatment group. | -7.00 (NA) — Only 1 participant evaluable in this treatment group. | -1.33 (2.082) | -1.27 (2.404)
  Change at Week 5 (Total Score): number analyzed (Participants) | 16 | 6 | 6 | 8 | 34
  Change at Week 5 (Total Score) | -8.88 (12.832) | -10.00 (7.616) | 5.33 (16.860) | 2.34 (12.010) | -4.21 (18.216)
  Change at Week 10 (Total Score): number analyzed (Participants) | 16 | 5 | 2 | 6 | 30
  Change at Week 10 (Total Score) | -8.75 (10.951) | -3.60 (8.649) | 6.50 (7.778) | 0.13 (10.569) | -11.40 (18.448)
  Change at Week 15 (Total Score): number analyzed (Participants) | 7 | 1 | 1 | 3 | 15
  Change at Week 15 (Total Score) | -7.86 (12.456) | 0.00 (NA) — Only 1 participant evaluable in this treatment group. | 13.00 (NA) — Only 1 participant evaluable in this treatment group. | -9.08 (13.135) | 0.73 (17.260)

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: The safety laboratory tests including Hematology, Clinical Chemistry and Urinalysis were performed.
  Determination if there were any laboratory data abnormalities of potential clinical concern was based on Pfizer Data Standards.
  Incidence of laboratory test abnormalities (without regard to baseline abnormality) was summarized within each treatment group.
Time Frame: Baseline (Day 0) to Week 17
Population: Safety Analysis Set included all participants who received at least 1 dose of PF-06649751 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
Participants | 19 | 4 | 9 | 7 | 25

8. Secondary Outcome: Number of Participants With Vital Sign Results Meeting the Criteria for Categorical Summarization
Description: Vital Signs including blood pressure and pulse rate were measured. Vital signs were collected first while the participant was in the supine position and then in the standing position.
Time Frame: Baseline (Day 0) to Week 17
Population: Safety Analysis Set included all participants who received at least 1 dose of PF-06649751 or placebo and had evaluable data at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 23 | 13 | 15 | 13 | 44
Participants
  <90 mmHg (Supine Systolic Blood Pressure [SBP]) | 1 | 1 | 2 | 0 | 3
  Max-Increase from Baseline >= 30 mmHg (Supine SBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Increase from Baseline >= 30 mmHg (Supine SBP) | 4 | 1 | 2 | 1 | 3
  Max-Decrease from Baseline >= 30 mmHg (Supine SBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Decrease from Baseline >= 30 mmHg (Supine SBP) | 4 | 1 | 2 | 2 | 11
  <90 mmHg (Standing SBP) | 4 | 1 | 3 | 2 | 7
  Max-Increase from Baseline >=30mmHg (Standing SBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Increase from Baseline >=30mmHg (Standing SBP) | 4 | 0 | 3 | 1 | 3
  Max-Decrease from Baseline >=30mmHg (Standing SBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Decrease from Baseline >=30mmHg (Standing SBP) | 3 | 0 | 3 | 2 | 12
  <50 mmHg (Supine Diastolic Blood Pressure [DBP]) | 0 | 0 | 0 | 1 | 1
  Max-Increase from Baseline >=20 mmHg (Supine DBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Increase from Baseline >=20 mmHg (Supine DBP) | 1 | 0 | 0 | 1 | 3
  Max-Decrease from Baseline >=20 mmHg (Supine DBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Decrease from Baseline >=20 mmHg (Supine DBP) | 1 | 0 | 2 | 1 | 13
  <50 mmHg (Standing DBP) | 2 | 0 | 1 | 2 | 1
  Max-Increase from Baseline >=20mmHg (Standing DBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Increase from Baseline >=20mmHg (Standing DBP) | 3 | 0 | 2 | 0 | 1
  Max-Decrease from Baseline >=20mmHg (Standing DBP): number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
  Max-Decrease from Baseline >=20mmHg (Standing DBP) | 5 | 2 | 3 | 2 | 17
  <40 beats per minute (bpm) (Supine Pulse Rate) | 0 | 0 | 0 | 0 | 0
  >120 bpm (Supine Pulse Rate) | 0 | 0 | 0 | 0 | 0
  <40 bpm (Standing Pulse Rate) | 0 | 0 | 0 | 0 | 0
  >140 bpm (Standing Pulse Rate) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Results Meeting the Criteria for Categorical Summarization
Description: The average of the triplicate readings of ECG data was collected at each assessment time.
  Number of participants with ECG results meeting the criteria for categorical summarization for time from the beginning of the P wave until the beginning of the QRS complex (PR Interval), time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization (QRS Duration), time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (QT Interval) and corrected QT (Fridericia correction) (QTcF Interval) were presented.
Time Frame: Baseline (Day 0) to Week 17
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 23 | 12 | 15 | 13 | 44
Participants
  >=300 msec (PR Interval) | 1 | 0 | 0 | 0 | 0
  Max-Increase From Baseline(%)>=25/50%(PR Interval): number analyzed (Participants) | 23 | 12 | 15 | 12 | 43
  Max-Increase From Baseline(%)>=25/50%(PR Interval) | 0 | 0 | 0 | 0 | 0
  >=140 msec (QRS Duration) | 0 | 0 | 0 | 0 | 0
  Max-Increase From Baseline(%)>=50% (QRS Duration): number analyzed (Participants) | 23 | 12 | 15 | 12 | 43
  Max-Increase From Baseline(%)>=50% (QRS Duration) | 0 | 0 | 0 | 0 | 0
  >=500 msec (QT Interval) | 1 | 0 | 0 | 0 | 0
  450 - <480 msec (QTcF Interval) | 2 | 0 | 0 | 0 | 1
  480 - <500 msec (QTcF Interval) | 0 | 0 | 0 | 0 | 0
  >=500 msec (QTcF Interval) | 0 | 0 | 0 | 0 | 0
  Max-Increase From Baseline 30-<60 (QTcF Interval): number analyzed (Participants) | 23 | 12 | 15 | 12 | 43
  Max-Increase From Baseline 30-<60 (QTcF Interval) | 1 | 0 | 0 | 0 | 1
  Max-Increase From Baseline >=60 (QTcF Interval): number analyzed (Participants) | 23 | 12 | 15 | 12 | 43
  Max-Increase From Baseline >=60 (QTcF Interval) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Suicidal Ideation Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) at Post-baseline Visits
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) was an interview based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS responses were mapped to the C-CASA. There were 3 key endpoints for suicidality data analysis and evaluation:
  * Suicidal Behavior: A participant was said to have suicidal behavior if the participant had experienced completed suicide / suicide attempt / reparatory acts toward imminent suicidal behavior.
  * Suicidal Ideation: Any observed suicidal ideation mapped to a single C-CASA category.
  * Suicidal Behavior or Ideation (participants with new onset suicidality): A participant was considered to have a new onset of suicidality if the participant reported no ideation and no behavior at the baseline assessment and reported any behavior or ideation post-baseline. Data observed at screening was not considered in the definition of worsening.
Time Frame: Days 0 (Baseline), 7, 14, 21, 28, 35, 70, 77, 84, 91, 105 and 119
Population: Safety Analysis Set included all participants who received at least 1 dose of PF-06649751 or placebo and had evaluable data at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 23 | 13 | 15 | 13 | 44
Participants
  Baseline | 1 | 0 | 1 | 0 | 0
  Day 7: number analyzed (Participants) | 22 | 11 | 14 | 12 | 44
  Day 7 | 0 | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 19 | 7 | 10 | 9 | 39
  Day 14 | 0 | 0 | 0 | 0 | 1
  Day 21: number analyzed (Participants) | 21 | 10 | 10 | 8 | 39
  Day 21 | 0 | 0 | 0 | 0 | 2
  Day 28: number analyzed (Participants) | 19 | 8 | 9 | 11 | 39
  Day 28 | 0 | 0 | 0 | 0 | 0
  Day 35: number analyzed (Participants) | 21 | 8 | 7 | 10 | 36
  Day 35 | 0 | 0 | 0 | 0 | 1
  Day 70: number analyzed (Participants) | 20 | 6 | 7 | 7 | 32
  Day 70 | 0 | 0 | 0 | 0 | 0
  Day 77: number analyzed (Participants) | 6 | 0 | 0 | 0 | 9
  Day 77 | 0 |  |  |  | 0
  Day 84: number analyzed (Participants) | 7 | 0 | 0 | 0 | 8
  Day 84 | 0 |  |  |  | 0
  Day 91: number analyzed (Participants) | 6 | 0 | 0 | 0 | 6
  Day 91 | 0 |  |  |  | 0
  Day 105: number analyzed (Participants) | 17 | 4 | 3 | 6 | 25
  Day 105 | 0 | 0 | 0 | 1 | 0
  Day 119: number analyzed (Participants) | 15 | 1 | 0 | 3 | 25
  Day 119 | 0 | 0 |  | 0 | 0

11. Secondary Outcome: Change From Baseline in Total Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease - Rating Scale (QUIP-RS)
Description: The QUIP-RS was a brief, patient reported outcome measure designed to assess the severity of symptoms of Impulsive-Compulsive Disorders (ICDs) and related behaviors reported to occur in Parkinson's disease.
  The QUIP-RS assessed 7 disorders (Gambling, Sex, Buying, Eating, Hobbyism-punding [performing tasks and repeating activities] and Taking medications). If more than 5 items were missing, the total QUIP-RS score was set as missing; otherwise, the total QUIP-RS score was imputed as follows: sum of the non-missing item scores * (total number of items) / (number of items non-missing). The higher score indicated a greater level of the ICD.
  The total QUIP-RS score for all ICDs and related disorders combined ranges from 0 to 112.
Time Frame: Baseline (Day 0) and Weeks 5, 10 and 15
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 23 | 13 | 15 | 13 | 44
units on a scale
  Baseline | 17.1 (16.98) | 9.0 (12.56) | 9.0 (14.39) | 12.5 (11.69) | 6.8 (11.40)
  Change at Week 5: number analyzed (Participants) | 22 | 11 | 10 | 12 | 42
  Change at Week 5 | -5.6 (11.37) | 2.3 (10.05) | 4.7 (9.58) | -5.4 (12.28) | 0.5 (11.13)
  Change at Week 10: number analyzed (Participants) | 20 | 5 | 6 | 6 | 30
  Change at Week 10 | -3.3 (12.16) | -1.8 (7.98) | -6.5 (9.63) | -5.8 (13.50) | 1.0 (10.62)
  Change at Week 15: number analyzed (Participants) | 16 | 4 | 3 | 4 | 24
  Change at Week 15 | -11.5 (16.29) | 3.0 (10.30) | -3.3 (5.77) | -17.0 (11.34) | 0.4 (5.91)

12. Secondary Outcome: Total Physician Withdrawal Checklist (PWC-20) on Days 105 and 119, and Change From Day 105 to Day 119
Description: The PWC-20 is a physician completed, 20 item reliable and sensitive instrument for the assessment of discontinuation symptoms. The PWC-20 was collected after the completion of study treatment and also at the first visit of follow-up.
  The total PWC-20 score was the sum of 20 item scores and ranged from 0 to 60. If more than 5 items were missing, the total PWC-20 score was missing; otherwise, the total PWC-20 score was imputed as follows: sum of the non-missing items * (total number of items) / (number of items non-missing). The higher score indicated more frequent/severe symptoms.
Time Frame: Days 105 and 119
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 23 | 13 | 15 | 13 | 44
units on a scale
  Day 105 Early Termination (ET): number analyzed (Participants) | 22 | 12 | 13 | 13 | 40
  Day 105 Early Termination (ET) | 3.5 (3.73) | 5.6 (5.68) | 5.8 (6.65) | 8.2 (8.78) | 7.1 (6.06)
  Day 119 Follow-up (FU): number analyzed (Participants) | 15 | 1 | 0 | 3 | 25
  Day 119 Follow-up (FU) | 3.3 (3.08) | 6.0 (NA) — Only 1 participant evaluable in this treatment group. |  | 7.7 (4.16) | 5.8 (5.45)
  Change From Day 105 ET to Day 119 FU: number analyzed (Participants) | 14 | 1 | 0 | 3 | 24
  Change From Day 105 ET to Day 119 FU | -0.6 (3.08) | -11.0 (NA) — Only 1 participant evaluable in this treatment group. |  | -1.7 (4.73) | -0.4 (4.79)

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Discontinuation Due to AEs and Deaths
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event did not need necessarily to have a causal relationship with the treatment or usage.
  An SAE was any untoward medical occurrence at any dose that:
  * Resulted in death;
  * Was life threatening (immediate risk of death);
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions);
  * Resulted in congenital anomaly/birth defect.
Time Frame: Day 1 to follow-up (Week 19 visit)
Population: Safety Analysis Set included all participants who received at least 1 dose of PF-06649751 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
Number analyzed (Participants) | 23 | 13 | 15 | 13 | 44
Participants
  AEs | 20 | 7 | 11 | 10 | 37
  SAEs | 1 | 1 | 0 | 0 | 2
  Discontinuation due to AEs | 3 | 1 | 3 | 2 | 9
  Death | 1 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to follow-up (Week 19 visit)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Placebo | PF-06649751 1 mg QD | PF-06649751 3 mg QD | PF-06649751 7 mg QD | PF-06649751 15 mg QD
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/13 | 0/15 | 0/13 | 1/44
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/13 | 0/15 | 0/13 | 2/44
Other Adverse Events (participants affected / at risk) | 15/23 | 7/13 | 11/15 | 10/13 | 31/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | PF-06649751 1 mg QD (N=13) | PF-06649751 3 mg QD (N=15) | PF-06649751 7 mg QD (N=13) | PF-06649751 15 mg QD (N=44)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic oedema (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | PF-06649751 1 mg QD (N=13) | PF-06649751 3 mg QD (N=15) | PF-06649751 7 mg QD (N=13) | PF-06649751 15 mg QD (N=44)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 11 (14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (3)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Dyskinesia (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 3 (3) | 7 (7)
Dystonia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 11 (14)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depersonalisation/derealisation disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysphemia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersexuality (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to insufficient efficacy and not due to safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT02687542/SAP_000.pdf
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT02687542/Prot_001.pdf